CLINICAL TRIAL: NCT02096315
Title: A Phase II, Open-label, Multicenter Study to Assess the Tolerance, Safety, Efficacy and Pharmacokinetics/Pharmacodynamics (PK/PD) of POL7080 in the Treatment of Patients With Acute Exacerbation of Non-cystic Fibrosis Bronchiectasis Due to Pseudomonas Aeruginosa Infection Requiring Intravenous Treatment
Brief Title: Safety, Efficacy and PK/PD of POL7080 in Patients With Exacerbation of Non-cystic Fibrosis Bronchiectasis.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Polyphor Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POL7080-002
Record Dates: First submitted 2014-03-18; First posted 2014-03-26 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2015-11

CONDITIONS: Bronchiectasis; Lower Respiratory Infection
Keywords: POL7080; Pseudomonas aeruginosa; Non cystic fibrosis bronchiectasis; Exacerbation
MeSH Terms: conditions — Bronchiectasis; Pseudomonas Infections | interventions — murepavadin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- POL7080 (Experimental): POL7080 administered daily
  Interventions: Drug: POL7080

INTERVENTIONS:
Drug: POL7080 — Intravenous infusion

SUMMARY:
To test whether POL7080 is effective in patients with exacerbation of non-cystic fibrosis bronchiectasis caused by Pseudomonas aeruginosa infection.

DETAILED DESCRIPTION:
* Patients will be recruited after written informed consent.
* Adverse events will be coded using Medical Dictionary for regulatory activities (MedDRA).
* Descriptive statistics will be used for all the safety and efficacy variables.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female aged ≥18 to <80 years and suffering from exacerbation of non-cystic fibrosis bronchiectasis due to Pseudomonas aeruginosa infection
2. Sputum sample collected for culture before starting treatment

Exclusion Criteria:

1. Female patients who are pregnant or breast feeding or unwilling to follow reliable method of contraception
2. Subjects suffering from cystic fibrosis, active pulmonary mycobacterial infection, end stage chronic obstructive pulmonary disease on long term oxygen therapy, severe uncontrolled asthma, active sarcoidosis and active allergic broncho-pulmonary aspergillosis
3. Current exacerbation of bronchiectasis is associated with lung abscess or empyema
4. Current exacerbation episode is suspected or documented to be due to pathogens other than Pseudomonas aeruginosa
5. Patients with known HIV infection with CD4+ (cluster of differentiation 4) cell count < 200/mm3
6. Patients who are currently enrolled in, or have not yet completed at least 30 days since ending another investigational device or drug trial or are receiving other investigational agent

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-12; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Sputum bacterial clearance | Day 4, Day 5, Day 10, Day 15 and Day 20
  Reduction in CFU/mL (colony forming units/mL) of Pseudomonas aeruginosa

SECONDARY OUTCOMES:
Adverse events | Daily assessment up to 20 days from informed consent.
  Number of adverse events reported by the patients or observed by the investigator will be recorded. Onset, end date, severity, causal relationship, outcome and measures taken will be summarized. Death, discontinuations and serious adverse events will be listed and narrative summaries will be provided.
Laboratory abnormalities. | Day 4, Day 10, Day 15 and Day 20
  The number and severity of abnormal blood chemistry and hematology findings will be summarized descriptively and compared to baseline. Clinically significant values/outliers will be listed and commented.
Volume of sputum in 24 hours | Day 4, Day 10, Day 15 and Day 20
  Reduction in 24 hours sputum volume as compared to baseline will be computed

OTHER OUTCOMES:
To measure the plasma concentrations of POL7080 | Day 3
  Blood samples to measure POL7080 concentrations before, during and after administration of POL7080

CONTACTS AND LOCATIONS:
Overall Officials: Eva Polverino, MD, Principal Investigator — Hospital Clinic, Barcelona, SPAIN; Adam Hill, MD PhD, Principal Investigator — Royal Infirmary, Edinburgh, U.K.
Locations (4):
- Spain (3):
  - Hospital Bellvitge, Barcelona
  - Hospital Clinic, Barcelona
  - Hospital La Fe, Valencia
- Royal Infirmary, City of Edinburgh, United Kingdom